CLINICAL TRIAL: NCT05991960
Title: Evaluation of Real-World Data on the Performance of the TECNIS Odyssey™ IOL
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DIOL112MRWD
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Intervention — No study treatments will be administered during this retrospective study. However, data will be collected from medical records of patients who have been treated with the subject device of this study.

SUMMARY:
Retrospective collection of data from medical records, multicenter, post-market clinical follow-up study.

ELIGIBILITY:
Inclusion Criteria:

1. Previously bilaterally implanted with TECNIS Odyssey IOL, following cataract extraction;
2. Enrollment at least 21 days after second eye surgery;
3. Clear intraocular media in each eye.
4. Signed consent and data protection documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries.

Exclusion Criteria:

1. Concurrent participation in an interventional clinical trial during the time from which the data will be collected;
2. Use of systemic or ocular medication that may affect vision;
3. Prior corneal refractive surgery in each eye (i.e., LASIK, PRK, SMILE, RK, CK); NOTE: Limbal relaxing incisions (LRI) are permissible as planned at the time of surgery (intraoperatively) but not postoperatively within the retrospective analysis window;
4. Ongoing adverse events in each eye that might impact outcomes during the study visit as determined by the investigator;
5. Acute or chronic disease or condition, ocular trauma or surgery that may affect vision in each eye (e.g., clinically significant macular degeneration, glaucoma, cystoid macular edema, proliferative diabetic retinopathy, keratoconus etc.).
6. Amblyopia, strabismus, nystagmus in each eye.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pseudophakic patients previously bilaterally implanted with TECNIS Odyssey IOL.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 1-month postoperative
  Visual Acuity will be collected via observed case data in units of logMAR.
Manifest Refraction | 1-month postoperative
  Manifest Refraction will be collected via observed case data in units of diopters.
Visual Symptoms/Complaints | 1-month postoperative
  Visual Symptoms/Complaints will be measured using a questionnaire on a 5-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision, Inc. Clinical Trial, Study Director — Johnson & Johnson Surgical Vision, Inc.
Locations (12):
- United States (12):
  - Assil Eye Institute, Beverly Hills, California
  - The Eye Institute of West Florida, Largo, Florida
  - Center for Sight, Sarasota, Florida
  - Aloha Vision Consultants, Honolulu, Hawaii
  - OCLI Vision, Garden City, New York
  - Vance Thompson Vision, West Fargo, North Dakota
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Carolina EyeCare Physicians, Mt. Pleasant, South Carolina
  - Loden Vision Centers, Goodlettsville, Tennessee
  - Dell Laser Consultants, Austin, Texas
  - Whitsett Vision Group, Houston, Texas
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu